CLINICAL TRIAL: NCT00855114
Title: A Phase II Trial of Short-Term Everolimus (RAD001) to Predict Response in Women With Operable Breast Cancer
Brief Title: Everolimus in Treating Women With Breast Cancer That Can Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to no accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS029; 0505M70026 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage III breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Treated with Everolimus (Experimental): Breast cancer patients treated with Everolimus by mouth, 5 mgs/day x 7 days, followed by surgery.
  Interventions: Drug: everolimus; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: everolimus — 5 mg/day x 7 days by mouth
  Other Names: RAD001; Afinitor(R)
Procedure: therapeutic conventional surgery — Definitive excision of breast cancer tissue
  Other Names: surgery

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating women with breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the administration of everolimus results in a decrease of total choline, a surrogate marker of response, in at least 30% of women with resectable breast cancer.

Secondary

* Determine whether tumors with activated mTOR signaling, as measured by phosphorylation of 4E-BP1 and activity of cap dependent translational complex, will identify those women responsive to everolimus.

OUTLINE: Patients receive oral everolimus once daily on days 1-7 in the absence of disease progression or unacceptable toxicity. Within 24 hours after completing everolimus, patients undergo surgery.

Tumor tissue samples are collected at baseline and during surgery for the analysis of mTOR targets (i.e., 4E-BP1, p70S6 kinase phosphorylation), Ki67, cleaved caspase 3, and activity of cap dependent translational complex by immunohistochemical assays. Patients also undergo MRI/MRS before and after everolimus therapy for total choline and glucose levels measurement.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer

  * Resectable disease
* Measurable disease, defined as a primary breast mass > 2.0 cm by breast imaging or clinical exam
* Planning to undergo surgical resection after neoadjuvant therapy
* Menopausal status not specified
* Eastern Clinical Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 9.0 g/dL
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* Intracranial disease
* Hormone receptor status not specified
* Obese (> 250 pounds)
* Immunosuppression from any cause (e.g., known HIV infection)
* History of severe asthma and/or allergies
* History of severe claustrophobia
* Ferromagnetic implants, history of shotgun wound and/or shrapnel, cardiac pacemakers, or other similar situations that would be contrary to strong magnetic force
* Bleeding diathesis
* Unstable systemic disease, including but not limited to, any of the following:

  * Uncontrolled diabetes
  * Severe infection
  * Severe malnutrition
  * Uncontrolled hypertension
  * Unstable angina
  * Ventricular arrhythmias
  * Active ischemic heart disease
  * Congestive heart failure
  * Myocardial infarction within the past 6 months
  * Chronic liver disease
  * Renal disease
  * Active upper gastrointestinal tract ulceration
* Less than 4 weeks since prior investigational drug
* Prior therapy with sirolimus or its analogues
* Concurrent immunosuppressive therapy (e.g., steroids, cytotoxic agents, or concurrent radiotherapy)
* Concurrent anticoagulation (i.e., coumadin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Decrease of total choline in at least 30% of patients | Pre-Treatment Compared to Post-Treatment (Day 7)
  Choline is measured by magnetic resonance imaging (MRI/MRS) scan.

SECONDARY OUTCOMES:
Identification of response to everolimus by activated mTOR signaling | Pre-Treatment Compared to Post-Surgery (Day 7)
  Two core biopsies will be obtained at the time of diagnostic biopsy. Waste tumor tissue obtained during surgery will be collected at the time of surgery. It will be stored under liquid nitrogen until they can be examined for activation of mTOR targets, specifically, 4E-BP1, p70S6 kinase phosphorylation, and activity of cap dependent translational complex.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Yee, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota, United States